CLINICAL TRIAL: NCT00673985
Title: A Randomized Study Comparing the Edwards Self-ExpandIng LifeStent Versus Angioplasty-alone In LEsions INvolving The SFA and/or Proximal Popliteal Arter
Brief Title: Edwards Lifesciences Self-Expanding Stent Peripheral Vascular Disease Study
Acronym: RESILIENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-12
Record Dates: First submitted 2008-02-14; First posted 2008-05-07 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Intermittent Claudication; Atherosclerotic Disease; Arterial Occlusive Disease
Keywords: SFA, Edwards, Popliteal, LifeStent, PTA, Nitinol
MeSH Terms: conditions — Intermittent Claudication; Arterial Occlusive Diseases; Truncus Arteriosus, Persistent | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): PTA Only: Active Comparator
  Percutaneous transluminal angioplasty (PTA) alone
  Interventions: Other: Percutaneous Transluminal Angioplasty
- 2 (Experimental): Test Arm: Experimental
  The main objective of this study is to assess the safety and effectiveness of the Edwards Lifesciences LifeStent nitinol self expandable stent device and its delivery system in the treatment of occlusive superficial femoral artery (SFA) disease.
  Interventions: Device: LifeStent NT™ Self-Expanding Peripheral Stent

INTERVENTIONS:
Other: Percutaneous Transluminal Angioplasty — Balloon Angioplasty
  Arms: 1
Device: LifeStent NT™ Self-Expanding Peripheral Stent — Balloon angioplasty plus stent
  Arms: 2

SUMMARY:
The main objective of this study is to assess the safety and effectiveness of the Edwards Lifesciences LifeStent nitinol self expandable stent device and its delivery system in the treatment of occlusive superficial femoral artery (SFA) disease by reducing the re-intervention rate as compared to percutaneous transluminal angioplasty (PTA) alone

DETAILED DESCRIPTION:
The RESILIENT Trial is a dual stage clinical investigation designed to evaluate the safety and effectiveness of the Edwards Lifesciences self-expanding stent system.

Phase 1 consists of a prospective, multi-center, non-randomized study with a peri-procedure endpoint. Phase 2 consists of a prospective, multi-center, randomized study with a 30-day primary safety endpoint and a 6-month primary effectiveness endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent approved by the IRB.
* ≥ 18 years old.
* Lifestyle-limiting claudication defined as: Rutherford Cat. 1-3.
* Target lesion(s) is de-novo or restenotic and located within the native SFA and/or proximal popliteal artery
* Angiographic evidence of ≥ 50% stenosis or occlusion
* Target RVD is ≥ 4.0 mm and ≤ 7.0 mm
* Target total length of the lesion or series of lesions is ≤ 150 mm.
* Angiographic evidence of at least one vessel runoff to the foot.

Exclusion Criteria:

* Unable to conform to the study protocol procedures and visits.
* Lifestyle-limiting claudication/CLI (Rutherford Cat. 4-6)
* Patients who are pregnant or planning to become pregnant during the clinical investigation
* Contraindication to study related medications, Ni, Ti, Ta, or other media that is not amenable to pretreatment.
* History of bleeding diatheses or coagulopathy.
* Concomitant renal failure with a creatinine of > 2.0 mg/dL.
* Concomitant hepatic insufficiency, thrombophlebitis, uremia, SLE, or DVT at the time of the study procedure.
* Receiving dialysis or immunosuppressive therapy.
* Suffered a hemorrhagic stroke ≤ 6 mo prior to the study procedure.
* Prior peripheral vascular bypass surgery involving the target limb.
* Target vessel has been previously stented.
* Target lesion(s) received angioplasty intervention ≤ 6 mo. prior
* Any non-iliac percutaneous intervention(s) < 7 days prior.
* Currently participating in an investigational drug/device study.
* Limited life expectancy of less than two years.
* Extensive PVD that precludes safe insertion of an sheath.
* Target lesion(s) is located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion(s).
* Unresolved thrombus within the target vessel.
* Poor inflow which would not support a vascular bypass graft.
* Diagnosed with septicemia at the time of the study procedure.
* Additional percutaneous interventional procedures (cardiac/peripheral) planned ≤ 30 days following procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2004-07; Primary Completion 2006-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety: Freedom from death at 30 days post-procedure. Effectiveness: Freedom from Target Lesion Revascularization (TLR) and/or Target Vessel Revascularization (TVR) at 6 months post-procedure. | 30 Day, 6 Month, and 12 Month

SECONDARY OUTCOMES:
Safety: Freedom from death, stroke, myocardial infarction, emergent surgical revascularization, significant distal embolization in target limb, and thrombosis of target vessel at 30-days post-procedure. Freedom from 30-day death and 6-month | 30 Day, 6 Month and12 Month

CONTACTS AND LOCATIONS:
Overall Officials: Barry T Katzen, MD, Principal Investigator — Baptist Cardiac & Vascular Institute, Miami, FL; John R Laird, MD, Principal Investigator — Vascular Center at the University of California, Davis Medical Center

REFERENCES:
- [Derived] Laird JR, Katzen BT, Scheinert D, Lammer J, Carpenter J, Buchbinder M, Dave R, Ansel G, Lansky A, Cristea E, Collins TJ, Goldstein J, Cao AY, Jaff MR; RESILIENT Investigators. Nitinol stent implantation vs. balloon angioplasty for lesions in the superficial femoral and proximal popliteal arteries of patients with claudication: three-year follow-up from the RESILIENT randomized trial. J Endovasc Ther. 2012 Feb;19(1):1-9. doi: 10.1583/11-3627.1. PMID 22313193
- [Derived] Laird JR, Katzen BT, Scheinert D, Lammer J, Carpenter J, Buchbinder M, Dave R, Ansel G, Lansky A, Cristea E, Collins TJ, Goldstein J, Jaff MR; RESILIENT Investigators. Nitinol stent implantation versus balloon angioplasty for lesions in the superficial femoral artery and proximal popliteal artery: twelve-month results from the RESILIENT randomized trial. Circ Cardiovasc Interv. 2010 Jun 1;3(3):267-76. doi: 10.1161/CIRCINTERVENTIONS.109.903468. Epub 2010 May 18. PMID 20484101